CLINICAL TRIAL: NCT00661297
Title: A Randomised, Double-blind, Parallel-group, Placebo-controlled Study Evaluating the Efficacy, Safety, and Reliability of 10mg Vardenafil Administered for 12 Weeks Compared to Placebo in Subjects With Erectile Dysfunction
Brief Title: Study Evaluating the Efficacy, Safety, and Reliability of Vardenafil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100536
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10 mg Vardenafil to be taken 1 h prior to sexual attempt
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
Study to investigate the efficacy and safety of Vardenafil

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual males
* >/= 18 years old with ED for more than six months
* Subjects also needed a positive first-time response to a single dose of 10mg vardenafil to be eligible for randomisation

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy
* Other exclusion criteria apply according to the Summary of Product Characteristics

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2003-06; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Sexual Encounter Profile question 2 (SEP 2) | 12 weeks

SECONDARY OUTCOMES:
Sexual Encounter Profile question 3 (SEP 3) | 12 weeks
International Index of Erectile Function (IIEF) - EF (Erectile Function) domain | 12 weeks
Safety and Tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer